CLINICAL TRIAL: NCT04947189
Title: 4CAST: A Phase 1b Dose Exploration and Dose Expansion, Open-label, Single-centre Study Evaluating the Safety and Efficacy of INO-464 in Combination With Chemotherapy in Patients With metASTatic Breast Cancer
Brief Title: Seviteronel in Combination With Chemotherapy in Androgen-receptor Positive Metastatic Triple-negative Breast Cancer
Acronym: 4CAST
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St Vincent's Hospital, Sydney (Other)
Responsible Party: Principal Investigator, Anthony Joshua, FRACP, Professor Anthony Joshua, St Vincent's Hospital, Sydney
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4CAST
Record Dates: First submitted 2021-03-25; First posted 2021-07-01 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Triple Negative Breast Cancer
Keywords: Androgen receptor positive
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Dexamethasone; seviteronel; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Seviteronel, dexamethasone and docetaxel (Experimental): Part 1: Seviteronel will be administered orally beginning with 450 mg (3 x 150 mg tablets) once daily along with 0.5 mg dexamethasone, continuously in 28-day cycles with docetaxel 75mg/m2 administered intravenously 3 weekly.
  Part 2: The recommended phase 2 dose for seviteronel (established in Part 1) once daily along with 0.5 mg dexamethasone, continuously in 21-day cycles with docetaxel 75mg/m2 administered intravenously 3 weekly.
  Interventions: Drug: Seviteronel-D (Seivteronel in combination with dexamethasone); Drug: Docetaxel

INTERVENTIONS:
Drug: Seviteronel-D (Seivteronel in combination with dexamethasone) — Use of Seviteronel-D (Serivteronel and dexamethasone) in the treatment of androgen receptor positive solid tumours.
  Other Names: INO-464
Drug: Docetaxel — Use of docetaxel chemotherapy for solid tumours

SUMMARY:
To facilitate the clinical testing of seviteronel and dexamethasone (SEVI-D) in combination with docetaxel in androgen receptor (AR) positive triple-negative breast cancer.

DETAILED DESCRIPTION:
Background:

Triple-negative breast cancer (TNBC) accounts for approximately 15-20% of all breast cancers and is defined by the absence of immunostaining for estrogen receptor (ER), progesterone receptor (PR), and non-amplified HER2 expression. Patients with metastatic TNBC exhibit a particularly poor clinical outcome, generally with rapid progression and a median overall survival (OS) rate of approximately 16 months. The current standard of care in the treatment of TNBC is cytotoxic chemotherapy and immunotherapy and the development of well-tolerated, effective, and targeted regimens that delay the need for cytotoxic chemotherapy and its side effects is an unmet need. Understanding breast cancer heterogeneity has enabled investigators to identify novel targets for the development of new therapeutic interventions. The androgen receptor (AR) is one such target. AR is expressed in 70-90% of all invasive breast cancers. Emerging data suggest that the AR-signalling pathway may play a critical role in breast cancer pathogenesis. Seviteronel is an orally bioavailable, selective cytochrome P450c17a (CYP17) lyase (lyase) and AR inhibitor. It is approximately 10-fold more selective for CYP17 lyase versus CYP17 17-α hydroxylase (hydroxylase) inhibition. Seviteronel inhibits the AR through competitive antagonism of both wild-type and mutated forms of the receptor. Through this unique, dual mechanism of action, it inhibits androgen production, thus reducing downstream estrogen aromatization from androgens, while also inhibiting AR binding and activation. In our own unpublished work, the investigators have shown that AR expression is often present in the cytoplasm of TNBC cells. When scoring patient samples for cytoplasmic AR, the investigators observed that ~cytoplasmic AR was present in 20% of TNBC patient tumours. This suggests that AR-targeted therapies may be beneficial for a far greater number of TNBC patients than is represented by the traditionally defined triple negative breast cancer AR subtype alone. Seviteronel has been shown to inhibit the growth in multiple breast cancer models, both in vitro and in vivo. Three early-phase prospective clinical studies investigating anti-androgen therapy have demonstrated clinical benefit of single-agent AR-targeted agents in women with metastatic AR positive TNBC. In our preliminary laboratory data (unpublished) demonstrates an increase in survival and suppression of metastatic TNBC when seviteronel is used in combination with docetaxel.

Aim:

To determine the feasibility, safety and efficacy of seviteronel and dexamethasone (SEVI-D) in combination with chemotherapy for the treatment of metastatic breast cancer. This study is conducted in two parts: part 1: dose exploration, and part 2: dose expansion.

Objectives:

To evaluate the safety and tolerability of SEVI-D and chemotherapy (docetaxel) in patients with metastatic breast cancer and determine the recommended phase II dose (RP2D) for SEVI-D/docetaxel combination therapy.

Part 1: Metastatic breast cancer

• To assess the pharmacokinetic and pharmacodynamic profiles of SEVI-D and chemotherapy (docetaxel) in metastatic breast cancer.

Part 2: Androgen receptor-positive metastatic triple-negative breast cancer

* To assess the pharmacokinetic and pharmacodynamic profiles of SEVI-D and chemotherapy (docetaxel).
* To evaluate the clinical activity SEVI-D and chemotherapy (docetaxel) in participants with cytoplasmic androgen receptor-positive metastatic triple negative breast cancer.

Design and sample size:

Part 1: Dose exploration - 6- 18 patients based on a rolling 6 design Part 2: Dose expansion - 35-45 patients in a single arm two-stage investigation

Study population:

Part 1: Patients with metastatic breast cancer. Part 2: Patients with cytoplasmic AR-positive metastatic triple-negative breast cancer confirmed by immunohistochemistry.

Study treatment:

Part 1: Seviteronel will be administered orally beginning with 450 mg (3 x 150 mg tablets) once daily along with 0.5 mg dexamethasone, continuously in 28-day cycles with docetaxel 75mg/m2 administered intravenously 3 weekly.

Part 2: The recommended phase 2 dose for seviteronel (established in Part 1) once daily along with 0.5 mg dexamethasone, continuously in 21-day cycles with docetaxel 75mg/m2 administered intravenously 3 weekly.

Screening for participation includes review of patient history, current health status, availability of a biospecimen for AR screening and patient willingness to be in a trial if eligible. Clinical and safety assessments are scheduled prior to registration and every 8 weeks until death. Imaging and other response assessments are required at baseline and every 2 cycles from cycle 1 day 1 until progression. Blood collection for translational studies will occur at: baseline (collected within 21 days prior to registration) or within 28 days of C1D1 treatment, every 2nd cycle and at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed written and voluntary informed consent.
* Patient must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
* Age 18 years or older male or female.
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* At least 4 weeks washout period from previous line of treatment, 2 weeks from radiotherapy
* Adequate haematologic and organ function within 14 days before the first study treatment on cycle1, day 1
* Life expectancy of at least 3 months
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods with a failure rate of <1% per year during the treatment period and for at least 28 days after the last dose of seviteronel or, 6 months after the last dose of chemotherapy whichever occurs later.
* Part 1: Histological or cytological-based diagnosis of breast cancer. Any of the three major subtypes of breast cancer is permitted for the phase 1b study, i.e., hormone receptor positive breast cancer i.e. oestrogen and/or progesterone positive in greater than 1% of cells by immunohistochemistry (IHC), or human epidermal growth factor receptor (HER2) positive breast cancer, i.e., IHC 3+ or in situ hybridisation (ISH) positive according to standard ASCO/CAP guidelines or triple-negative breast cancer, i.e., HER2-negative by ASCO/GAO Guidelines and <1% expression of estrogen and/or progesterone receptor by IHC.
* Part 2: Histological or cytological-based diagnosis of triple-negative breast cancer. The tumor must be HER2-negative by ASCO/GAO Guidelines and <1% expression of estrogen and /or progesterone receptor by IHC.

  o The tumor must also show androgen receptor positivity (i.e., AR>0%) by IHC or gene classifier (molecular testing).
* Measurability of lesion: have at least 1 measurable lesion assessable using standard techniques by RECIST v1.1
* Patients must have advanced or recurrent breast cancer pre-inclusion number 8, for whom docetaxel is considered an appropriate treatment option.

Exclusion Criteria:

* Inability to comply with study and follow-up procedures.
* History of malabsorption syndrome or other condition that would interfere with enteral absorption or results in the inability or unwillingness to swallow pills.
* Active infection requiring antibiotics.
* Other invasive malignancy within 2 years except for malignancies determined to have low recurrence potential in discussion with study PI.
* Known active tuberculosis.
* Female patients who are pregnant or breast-feeding.
* Male or female patients of reproductive potential who are not willing to use effective birth control from screening to 90 days post treatment.
* Women of childbearing potential (who are not postmenopausal within 12 months of non-therapy induced amenorrhea, nor surgically sterile) must have a negative serum pregnancy test result within 3 days prior to initiation of study treatment.
* Uncontrolled intercurrent illness, including psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events, or compromise the ability of the subject to give written informed consent.
* History or current evidence of HIV infection.
* Known clinically significant history of liver disease consistent with Child-Pugh Class B or C, including active viral or other hepatitis (e.g., positive for hepatitis B surface antigen [HBsAg] or hepatitis C virus [HCV] antibody at screening), current drug or alcohol abuse, or cirrhosis:
* Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen antibody test) are eligible.
* Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 of Cycle 1 or anticipation of need for a major surgical procedure during the course of the study
* Placement of a vascular access device is not considered major surgery.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Patients with symptomatic central nervous system (CNS) metastasis and/or carcinomatous meningitis. Patients with treated CNS metastases are eligible for this study if they are not receiving corticosteroids and/or anticonvulsants for at least 7 days prior to first dose of study treatment, and their disease is asymptomatic and radiographically stable for at least 30 days prior to consent by repeat imaging (repeat imaging should be performed during study screening).
* Unresolved, clinically significant toxicity NCI CTCAE v5.0 grade 2 or higher, from prior therapy, except for alopecia, endocrinopathy on stable hormonal replacement, and others as approved by study PI.
* Patients who have received palliative radiation treatment to peripheral sites (e.g., bone metastases) for pain control and whose last treatment was completed 14 days prior to Day 1 of Cycle 1 may be enrolled in the study if they have recovered from all acute, reversible effects.
* Uncontrolled pleural effusion, pericardial effusion, or ascites.
* Known hypersensitivity or contraindication to any component of the study treatment.
* Administration of any investigational treatment within 30 days or 5 half-lives (whichever is longer) prior to receiving the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose of seviteronel plus dexamethasone and docetaxel | 10 weeks
  A patient will be considered evaluable for dose limiting toxicity (DLT) if they have completed two cycles of docetaxel in an 8-week period with at least 80% of the planned INO-464 dose. Toxicity will be graded using CTCAE version 5.0

SECONDARY OUTCOMES:
Number of patients with treatment-related adverse events | 2 years
  Incidence, nature, and severity of adverse events and laboratory abnormalities, with severity determined according to NCI CTCAE v5.0
Overall response rate (ORR) | 2 years
  The proportion of patients with a confirmed complete response or partial response as determined by the investigator according to RECIST v1.1
Duration of response (DoR) | 2 years
  The time from the first occurrence of a documented confirmed complete response or partial response to the first date of recorded disease progression, as determined by the investigator according to RECIST v1.1, or death from any cause (whichever occurs first)
Overall survival (OS) | 2 years
  The time from starting the study treatment to death from any cause

OTHER OUTCOMES:
Gene expression signatures in tumour biopsies treated with seviteronel | 2 years
  Gene expression analysis (RNAseq, or single-cell RNAseq) on tumor biopsies in response to study treatments.
Androgen receptor protein signature in biopsies treated with seviteronel | 2 years
  Expression of androgen receptor, ZEB1 and other protein markers in tumor biopsies in response to study treatment
Biomarker expression in blood and/or tumor tissue following seviteronel treatment | 2 years
  Gene expression and/or ctDNA analysis in blood and/or tumour biopsies in response to the study treatments.

CONTACTS AND LOCATIONS:
Locations (1):
- Kinghorn Cancer Centre, Darlinghurst, New South Wales, Australia